CLINICAL TRIAL: NCT03218683
Title: A Phase 1/1b/2a, 3-Part, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of Ascending Doses of AZD5991 Monotherapy and in Combination With Venetoclax in Subjects With Relapsed or Refractory Haematologic Malignancies
Brief Title: Study of AZD5991 Alone or in Combination With Venetoclax in Relapsed or Refractory Haematologic Malignancies.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6910C00001
Record Dates: First submitted 2017-07-06; First posted 2017-07-14 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia (AML)
Keywords: relapsed; refractory; AZD5991; Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — AZD5991; venetoclax

STUDY DESIGN:
Intervention Model Description: This study is a 3 part, multicenter, open-label, nonrandomized, sequential group, dose-escalation study to assess safety, tolerability,pharmacokinetics and preliminary anti-tumor activity of ascending doses of AZD5991 alone or in combination with venetoclax in subjects with relapsed or refractory hematologic malignancies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Monotherapy AZD5991 (Experimental): Dose escalation - multiple dose levels
  Interventions: Drug: AZD5991
- Monotherapy AZD5991 expansion (Experimental): Dose expansion
  Interventions: Drug: AZD5991
- AZD5991 + venetoclax (Experimental): Dose escalation - multiple dose levels
  Interventions: Drug: AZD5991 + Venetoclax

INTERVENTIONS:
Drug: AZD5991 — AZD5991 will be administered intravenously for 9 cycles (each cycle 21 days) or until patient derives treatment benefit or progresses
  Arms: Monotherapy AZD5991; Monotherapy AZD5991 expansion
Drug: AZD5991 + Venetoclax — Ascending oral doses of AZD5991 and/or venetoclax until no longer tolerated or disease progression
  Arms: AZD5991 + venetoclax

SUMMARY:
This study is a multicenter, open-label, nonrandomized, sequential group, dose-escalation study to assess safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of ascending doses of AZD5991 in subjects with relapsed or refractory hematologic malignancies Part 1 of the study is monotherapy dose escalation. Closed November 2020 Part 2 of the study is monotherapy expansion groups for relapsed/refractory chronic lymphocytic leukaemia (CLL), AML/ myelodysplastic syndromes (MDS), and multiple myeloma (MM). Closed November 2020 Part 3 is a sequential, dose-escalation study of the combination of AZD5991 and venetoclax in subjects with relapsed/refractory AML

ELIGIBILITY:
Inclusion Criteria (AZD5991 + venetoclax):

* Provision of signed and dated, written informed consent prior to any study-specific procedures, sampling and analyses.
* Men and women 18 to 85 years of age, inclusive.
* Diagnosis of AML and histologically proven based on criteria established by the World Health Organisation (WHO) as documented by medical records. Must have a measurable blast infiltration in bone marrow which will serve as a response parameter
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Must have received at least 1 prior line of therapy and there must be no treatment options available known to provide clinical benefit. Refer to National Comprehensive Cancer Network (NCCN) guidelines.
* Documented active disease requiring treatment per respective NCCN guideline that is relapsed or refractory defined as:
* Recurrence of disease after response to prior line(s) of therapy.
* Or progressive disease after completion of the treatment regimen preceding entry into the study.
* WBC ≤10,000 cells/mm3 (10 x 109/L); use of leukapheresis or hydroxyurea before study drug initiation is allowed to achieve this entry criterion.
* Adequate hepatic and renal function at screening defined as:
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 x upper limit of normal (ULN).
* Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin).
* Serum creatinine ≤1.5 times ULN and creatinine clearance ≥50 mL/min (measured or calculated by Cockcroft and Gault equation [(140-Age) • Mass (kg)/(72 • creatinine mg/dL) • multiply by 0.85 if female]).
* Lipase ≤1.5 x ULN and serum amylase ≤1.5 x ULN and no history of pancreatitis.
* Women should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test before start of dosing if of child-bearing potential or must have evidence of nonchildbearing potential.
* Men should be willing to use barrier contraception (ie, condoms) and refrain from sperm donation during and after the conduct of the trial.

Exclusion Criteria (AZD5991 + venetoclax):

* Treatment with any of the following:

  * Any investigational agents from a previous clinical study within 4 half-lives or 14 days, whichever is the greater, of said prior investigational agent(s) with regard to the first dose of study treatment on this protocol. Washout period not required in subjects with aggressive disease who require treatment sooner.
  * Any other chemotherapy, immunotherapy or anticancer agents within 2 weeks of the first dose of study treatment. Washout period not required in subjects with aggressive disease who require treatment sooner.
  * Any hematopoietic growth factors (eg, filgrastim [granulocyte colony-stimulating factor; G-CSF], sargramostin [granulocyte-macrophage colony-stimulating factor; GM-CSF]) within 7 days of the first dose of study drug or pegylated G-CSF (pegfilgrastim) or darbepoetin within 14 days of the first dose of study drug.
  * Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment.
* Except for alopecia, any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment.
* AML with known active central nervous system involvement.
* As judged by the Investigator, any evidence of severe or uncontrolled systemic disease (eg, severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease]), or current unstable or uncompensated respiratory or cardiac conditions, or uncontrolled hypertension, history of, or active, bleeding diatheses (eg, hemophilia or von Willebrand disease) or uncontrolled active systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment), or intravenous anti-infective treatment within 2 weeks before first dose of study drug.
* Malabsorption syndrome or other condition that precludes enteral route of administration.
* Chronic respiratory disease that requires continuous oxygen use.
* Known diagnosis of a hypercoagulable disorder other than malignancy
* Undergone any of the following procedures or experienced any of the following conditions currently or in the preceding 6 months:

  * angina pectoris
  * supraventricular arrhythmias, including atrial fibrillation, which are uncontrolled
  * Myocarditis
  * heart failure NYHA Class I or above
* Experienced any of the following conditions currently or at any previous timepoint

  * Myocardial infarction (MI)
  * coronary artery bypass graft
  * angioplasty
  * vascular stent
  * Heart failure NYHA Class ≥ 2
  * Ventricular arrhythmias requiring continuous therapy
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTcF) ≥ 450 msec applicable to both genders obtained from 3 electrocardiograms (ECGs) (averaged)
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, second to third degree AV block, sinus node dysfunction with clinically significant sinus pause
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age. Concomitant medications known to prolong QTc should be used with caution and cannot be used starting with the first dose of study drug and through the DLT review period.
  * ST-wave depression and T-wave changes (e.g. inversion or flattened) in recent or screening ECG
  * CPK assay reading ≥ ULN at screening
  * Subjects with any troponin assay reading of ≥ULN during screening
  * Left ventricular ejection fraction [LVEF] <55% with echocardiogram (ECHO) or multi-gated acquisition scan (MUGA). Appropriate correction to be used, if a MUGA is performed.
* History of severe allergic or anaphylactic reactions to BH3 mimetics or history of hypersensitivity to active or inactive excipients of AZD5991.
* Received the following within 7 days before initiation of venetoclax:
* Strong or moderate cytochrome P450 3A (CYP3A) inducers
* Strong or moderate CYP3A inhibitors
* Pg-P inhibitors
* Consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or star fruit within 3 days before the initiation of venetoclax.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | At every treatment and follow up visit until disease progression. Expected to be for up to 12 months
  Number of subjects with adverse events as a measure of safety and tolerability including changes in vital signs, electrocardiograms (ECGs), safety and laboratory parameters
Dose limiting toxicities | Minimum observation period is 28 days per cohort
maximum tolerated dose | Minimum observation period is 28 days for the maximum dose cohort

SECONDARY OUTCOMES:
Maximum observed plasma concentration of AZD5991 monotherapy and AZD5991+venetoclax | Predose and through 24 hours postdose
  To assess the pharmacokinetics of AZD5991 monotherapy and AZD5991+venetoclax
Area under the concentration-time curve for plasma concentrations of AZD5991 monotherapy and AZD5991+venetoclax | Predose and through 24 hours postdose
  To assess the pharmacokinetics of AZD5991 monotherapy and AZD5991+venetoclax
Objective response rate (ORR) | From time of first dose until discontinuation of AZD5991 monotherapy and AZD5991+venetoclax expected to be for up to 12 months
  To assess the antitumor activity of AZD5991 monotherapy and AZD5991+venetoclax. Response will be evaluated every 8-12 weeks during treatment until progression.
Duration of response (DOR) | From time of first dose until discontinuation of AZD5991 monotherapy and AZD5991+venetoclax expected to be for up to 12 months
  To assess the antitumor activity of AZD5991 monotherapy and AZD5991+venetoclax. Response will be evaluated every 8-12 weeks during treatment until progression.
Progression-free survival (PFS) | From time of first dose until first observation of progression expected to be for up to 12 months
  To assess the antitumor activity of AZD5991 monotherapy and AZD5991+venetoclax. Response will be evaluated every 8-12 weeks during treatment until progression.
Complete remission rate (CRR) | From time of first dose until discontinuation of AZD5991 monotherapy and AZD5991+venetoclax expected to be for up to 12 months
  To assess the antitumor activity of AZD5991 monotherapy and AZD5991+venetoclax. Response will be evaluated every 8-12 weeks during treatment until progression.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Research Site, Orange, California
  - Research Site, Aurora, Colorado
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] White MJ, Cheatham L, Wen S, Scarfe G, Cidado J, Reimer C, Hariparsad N, Jones RDO, Drew L, McGinnity DF, Vasalou C. A PKPD Case Study: Achieving Clinically Relevant Exposures of AZD5991 in Oncology Mouse Models. AAPS J. 2023 Jun 28;25(4):66. doi: 10.1208/s12248-023-00836-z. PMID 37380821
- [Derived] Tron AE, Belmonte MA, Adam A, Aquila BM, Boise LH, Chiarparin E, Cidado J, Embrey KJ, Gangl E, Gibbons FD, Gregory GP, Hargreaves D, Hendricks JA, Johannes JW, Johnstone RW, Kazmirski SL, Kettle JG, Lamb ML, Matulis SM, Nooka AK, Packer MJ, Peng B, Rawlins PB, Robbins DW, Schuller AG, Su N, Yang W, Ye Q, Zheng X, Secrist JP, Clark EA, Wilson DM, Fawell SE, Hird AW. Discovery of Mcl-1-specific inhibitor AZD5991 and preclinical activity in multiple myeloma and acute myeloid leukemia. Nat Commun. 2018 Dec 17;9(1):5341. doi: 10.1038/s41467-018-07551-w. PMID 30559424